CLINICAL TRIAL: NCT05764915
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of RGT-264 Phosphate Tablets in Subjects With Advanced Solid Tumors
Brief Title: A Phase I Study of RGT-264 in Subjects With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to the change in study plan and not due to safety reasons
Sponsor: Regor Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RGT-264-101; CTR20223017 (Other: CDE)
Record Dates: First submitted 2023-01-11; First posted 2023-03-13 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Advanced Solid Tumor
Keywords: Hematopoietic progenitor kinase 1 (HPK1); Dose Escalation; Dose Expansion; RGT-264; First-in-Human
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Intervention Model Description: There will be one arm in the study. Enrolled subjects will be treated with RGT-264 phosphate tablets alone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RGT-264 monotherapy (Experimental): The study is composed of dose escalation stage and dose expansion stage. RGT-264 will be administered orally daily alone as monotherapy in both stages. In the dose escalation stage, the subjects will receive once daily of RGT-264 monotherapy across approximately 6 ascending dose levels. The starting dose is 10 mg/day. In the dose expansion stage, the subjects will receive RGT-264 treatment at the recommended dose from dose escalation part.
  Interventions: Drug: RGT-264 phosphate tablets

INTERVENTIONS:
Drug: RGT-264 phosphate tablets — RGT-264 phosphate tablets will be administered orally once daily (QD).

SUMMARY:
This is a Phase 1 dose escalation and dose expansion study to evaluate the safety, tolerability, pharmacokinetics, and preliminary efficacy of RGT-264 as monotherapy in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
This first-in-human (FIH) study of RGT-264 will evaluate safety, pharmacokinetics (PK) and efficacy of RGT-264 in subjects with advanced solid tumors. The primary objective is to determine the maximum tolerated dose (MTD)/maximum administered dose (MAD) and the recommended phase II dose (RP2D) of RGT-264 as monotherapy, and to evaluate the safety and tolerability of RGT-264. The secondary objectives include the assessments of PK profile and preliminary efficacy of RGT-264.

ELIGIBILITY:
Inclusion Criteria:

* Able to sign the ICF and agree to comply with the requirements of the study;
* Subjects with pathologically confirmed advanced solid tumors who have failed standard-of-care therapy, or have no standard-of-care therapy available, or are currently not eligible for standard-of-care therapy;
* ECOG performance status score of 0 to 1;
* Expected survival ≥ 3 months;
* With at least one measurable lesion per RECIST v1.1;
* Subjects should discontinue all anti-tumor therapies prior to receiving study treatment, and the toxicity caused by prior anti-tumor therapy has recovered to ≤ Grade 1 per CTCAE v5.0;
* The specific requirements of washout period should be met before first dose;
* Adequate organ function
* Female subjects of childbearing potential must have a negative pregnancy test prior to the first dose and are required to use effective contraception from signing the ICF until 6 months after the last dose of study treatment

Exclusion Criteria:

* Presence of risks that may significantly affect the absorption of the investigational product (e.g. inability to swallow, intestinal obstruction, chronic diarrhea, etc.);
* Having received immunotherapy and experienced ≥ Grade 3 immune-related adverse events (irAEs) or ≥ Grade 2 immune-related myocarditis;
* Having received systemic glucocorticoids (> 10 mg/day of prednisone or equivalent) or other immunosuppressants within 14 days prior to the first dose of investigational product;
* Presence of symptomatic parenchymal brain metastasis or leptomeningeal metastasis;
* Active, or previous autoimmune disease with the potential for relapse (excluding well-controlled type 1 diabetes mellitus; manageable hypothyroidism with hormone replacement therapy only).;
* Any other malignancy (except cured basal cell carcinoma of skin and in-situ carcinoma of the cervix) within 3 years prior to the first dose;
* History of serious cardiovascular and cerebrovascular diseases;
* Presence of active interstitial lung disease or history of interstitial lung disease requiring glucocorticoid treatment;
* Presence of severe chronic or active infections (including tuberculosis infection, etc.) requiring intravenous antimicrobial, antifungal or antiviral therapy;
* Active HBV or HCV infection;
* History of immunodeficiency or organ transplantation;
* Presence of uncontrolled third spacing fluid;
* Concomitant diseases or any other conditions that may seriously jeopardize the subject's safety or affect the subject's completion of the study, at the discretion of the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Number of subjects with Dose-Limiting Toxicities (DLTs) at each cohort dose level in dose escalation stage | Day 1 to Day 21 after first dose (21 days)
  DLTs will be evaluated from Day 1 (the day of the first dose) to Day 21 after first dose of study treatment in escalation stage. Number of DLTs will be used in dose ascending and descending decisions.
Number of subjects with adverse events (AEs) | From screening (Day -28 to Day -1) through up to 12 months or until disease progression
  AEs will be characterized by type, seriousness, relationship to study treatment, severity (as graded by National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] version 5.0) and timing.

SECONDARY OUTCOMES:
Pharmacokinetic Assessments: Time to maximum plasma concentration (Tmax) | PK Blood (Cycle 1 Day 1 and Cycle 1 Day 15; PK Urine (Cycle 1 Day 1) (each cycle is 21 days)
  Blood and urine samples will be collected for PK analyses for subjects enrolled in dose escalation stage.
Pharmacokinetic Assessments: Maximum concentration (Cmax) | PK Blood (Cycle 1 Day 1 and Cycle 1 Day 15; PK Urine (Cycle 1 Day 1) (each cycle is 21 days)
  Blood and urine samples will be collected for PK analyses for subjects enrolled in dose escalation stage.
Pharmacokinetic Assessments: Elimination half-life (t1/2) | PK Blood (Cycle 1 Day 1 and Cycle 1 Day 15; PK Urine (Cycle 1 Day 1) (each cycle is 21 days)
  Blood and urine samples will be collected for PK analyses for subjects enrolled in dose escalation stage.
Pharmacokinetic Assessments: Area under the concentration-time curve over time 0 to t (AUC0-t) | PK Blood (Cycle 1 Day 1 and Cycle 1 Day 15; PK Urine (Cycle 1 Day 1) (each cycle is 21 days)
  Blood and urine samples will be collected for PK analyses for subjects enrolled in dose escalation stage.
Pharmacokinetic Assessments: Area under the concentration-time curve over time 0 to infinite (AUC0-inf) | PK Blood (Cycle 1 Day 1 and Cycle 1 Day 15; PK Urine (Cycle 1 Day 1) (each cycle is 21 days)
  Blood and urine samples will be collected for PK analyses for subjects enrolled in dose escalation stage.
Pharmacokinetic Assessments: Accumulation ratio (Rac) | PK Blood (Cycle 1 Day 1 and Cycle 1 Day 15; PK Urine (Cycle 1 Day 1) (each cycle is 21 days)
  Blood and urine samples will be collected for PK analyses for subjects enrolled in dose escalation stage.
Pharmacokinetic Assessments: Cumulative urinary excretion | Cycle 1 Day 1 (each cycle is 21 days)
  Urine samples will be collected for PK analyses for subjects enrolled in dose escalation stage.
Tumor Response | Screening until disease progression, initiation of a new anti-tumor therapy, death, loss to follow-up, withdrawal of consent, or meeting other end-of-study criteria (whichever occurs first) (Assessed up to 12 months).
  Tumor response measured by radiologic imaging techniques at baseline and throughout the study. The same radiologic imaging techniques for each respective patient will be used throughout. Tumor response will be assessed by investigator according to RECIST v1.1.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The First Affiliated Hospital Of Nanchang University City, Nanchang, Jiangxi
  - Shandong Provincial Institute of Cancer Prevention and Treatment, Jinan, Shandong
  - Shanghai East Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No